CLINICAL TRIAL: NCT02325661
Title: Open Uncontrolled Validation Study for the German Version of the Actinic Keratosis Quality of Life Questionnaire (AKQoL)
Acronym: AKQOLVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: KEK-ZH-Nr. 2014-0252
Record Dates: First submitted 2014-12-15; First posted 2014-12-25 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cognitive interviewing (Other): individual cognitive interviewing, 30 minutes per patient
  Interventions: Other: cognitive interviewing

INTERVENTIONS:
Other: cognitive interviewing — For the individual cognitive interviews we are using the two techniques "to think aloud" and the "verbal probing". "To think aloud" means, that the patients are asked to express precisely what comes to their mind when reading the single questions. This means, the interviewer is interested in the line of thoughts, which arise when reading the question. Thereby, the problems which appear in the usually covert process of answering a question should be revealed. In a second step, we are using the "verbal probing" technique to identify possible misunderstandings of the questions or difficulties with single phrases. The interviewer asks further questions that target the patients' interpretation.

SUMMARY:
The objective of this study is to translate the "AKQoL"-questionnaire which measures the quality of life of patients with actinic keratosis into German and to validate it for the Swiss population.

By using the technique of cognitive interviewing the investigators are focussing on the patients' understanding of the questions. The first session of cognitive interviews will show, where there is need for improvement in terms of misinterpreted phrases or vaguely worded questions. The goal is to rephrase the questions according to the feedback of the patients. The revised version will then be presented to a new population.

DETAILED DESCRIPTION:
Actinic keratosis is a UV-induced skin disease, which presents as a reddish, squamous and sometimes itchy lesion. Actinic keratosis seems to have a negative impact on patients' quality of life. Esmann et al. elaborated on patients with actinic keratosis from Zealand, Denmark a questionnaire which measures the quality of life.

The objective of this study is to translate this questionnaire into German and to validate it for the Swiss population. This questionnaire might become part of a planned national register for data collection of patients with AK.

The investigators will assess the content validity of the questionnaire by using the technique of cognitive interviewing. The investigators are going to talk 34 patients with AK from the department of Dermatology, University Hospital Zurich through the translated version. Thereby, the investigators are focusing on the patients' understanding of the questions.

The first session of cognitive interviews will show, where there is need for improvement in terms of misinterpreted phrases or vaguely worded questions. The goal is to rephrase the questions in the sense that they become more clear and are understood by different interviewee in the same way. The revised version will then be presented to a new population. The performance of cognitive interview sessions and revisions will continue until the survey will be approved by at least 80% of the respondents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with actinic keratosis of the department of Dermatology, University Hospital Zurich
* Male and Female subjects > 18 years of age
* Good understanding of written and spoken German
* Sufficient physical and mental capacity to comprehend the questions
* Written informed consent by the participant

Exclusion Criteria:

* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Intersubject agreement on validation of the questions of the AKQoL | 30 minutes per patient
  Consistent answers by study participants on cognitive debriefing. This is a qualitative, not a quantitative measure.

CONTACTS AND LOCATIONS:
Overall Officials: Günther Hofbauer, Prof.Dr.med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Esmann S, Vinding GR, Christensen KB, Jemec GB. Assessing the influence of actinic keratosis on patients' quality of life: the AKQoL questionnaire. Br J Dermatol. 2013 Feb;168(2):277-83. doi: 10.1111/bjd.12036. PMID 22962980